CLINICAL TRIAL: NCT03934632
Title: The Impact of Leg Immobilization on Postabsorptive and Postprandial Muscle Protein Breakdown in Healthy Young Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 180509/B/01
Record Dates: First submitted 2019-04-16; First posted 2019-05-02 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Healthy
MeSH Terms: interventions — Postprandial Period; Immobilization

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postabsorptive (Active Comparator): Saline infusion to mimic postabsorptive circulating amino acid concentrations
  Interventions: Other: Postabsorptive; Procedure: Immobilisation
- Postprandial (Active Comparator): Amino acid infusion to mimic postprandial circulating amino acid concentrations
  Interventions: Other: Postprandial; Procedure: Immobilisation

INTERVENTIONS:
Other: Postabsorptive — Saline will be infused to mimic postabsorptive circulating amino acid concentrations
  Arms: Postabsorptive
Other: Postprandial — An amino acid infusate will be administered to mimic postprandial circulating amino acid concentrations
  Arms: Postprandial
Procedure: Immobilisation — One leg will undergo 2 days immobilisation prior to the test day

SUMMARY:
The present study will seek the quantify the simultaneous muscle protein synthesis and breakdown response with and without amino acid provision in humans following 2 days of immobilisation.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-40 years of age
* Body mass index between 18.5 and 30

Exclusion Criteria:

* Any diagnosed metabolic impairment (e.g. type 1 or 2 Diabetes)
* Any diagnosed cardiovascular disease (e.g. deep vein thrombosis) or hypertension
* Chronic use of any prescribed or over the counter pharmaceuticals (that may modulate muscle protein metabolism)
* A personal or family history of epilepsy, seizures or schizophrenia
* Any known disorders in muscle metabolism
* Regular use of nutritional supplements
* Allergy to lidocaine
* Allergy to one or multiple amino acids
* Recent (within the last 6 months) or current musculoskeletal injury (e.g. leg fracture) as these could be exacerbated by the intervention e.g. unilateral leg immobilisation, or mean the participant is unable to use crutches.
* Having received or ingested a stable isotope tracer in the past

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Muscle protein breakdown rate | 1 hour
  Muscle protein breakdown rate (FBR, measured in %/h) during 1 hour of saline or amino acid infusion

SECONDARY OUTCOMES:
Muscle protein breakdown rate | 3 hours
  Muscle protein breakdown rate (FBR, measured in %/h) during 3 hours of saline or amino acid infusion
Muscle protein synthesis rate | 3 hours
  Muscle protein synthesis rate (FSR, measured in %/h) during 3 hours of saline or amino acid infusion measured using a D5 phenylalanine infusion

CONTACTS AND LOCATIONS:
Overall Officials: Marlou Dirks, PhD, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom